CLINICAL TRIAL: NCT02760121
Title: The Effect of Carbonic Anhydrase Inhibitors on the Pulmonary System Response to Hypoxia
Brief Title: AZ, MZ, and the Pulmonary System Response to Hypoxia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H16-00028
Record Dates: First submitted 2016-04-20; First posted 2016-05-03 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Altitude Sickness; Hypertension, Pulmonary
Keywords: Acetazolamide; Methazolamide; Control of breathing; Hypoxic pulmonary vasoconstriction
MeSH Terms: conditions — Altitude Sickness; Hypertension, Pulmonary | interventions — Acetazolamide; Methazolamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Acetazolamide (Experimental): Participants will be dosed 250mg Acetazolamide (p.o.) three times per day for two days prior to and a single dose on the day of study.
  Interventions: Drug: Acetazolamide
- Methazolamide (Experimental): Participants will be dosed 100mg Methazolamide (p.o.) twice daily separated by a placebo for two days prior to and a single dose on the day of study. The placebo dose is provided to match the dosing schedule between conditions.
  Interventions: Drug: Methazolamide
- Placebo (Placebo Comparator): Participants will take (p.o.) placebo pills three times per day for two days prior to and a single dose on the day of study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetazolamide
  Arms: Acetazolamide
Drug: Methazolamide
  Arms: Methazolamide
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this proposal is to compare the physiological effects of acetazolamide (AZ) and methazolamide (MZ) on the control of breathing and hypoxic pulmonary vasoconstriction. The first objective is to assess the effects of AZ and MZ on the control of breathing in normoxia and hypoxia. To achieve this the ventilatory interaction between oxygen and carbon dioxide will be measured and effects compared between placebo, AZ, and MZ conditions. In addition, the isocapnic and poikilocapnic hypoxic ventilatory response and hypercapnic ventilatory response will be measured with each drug. The second objective is to assess the effects of AZ and MZ on the control of the pulmonary vasculature during hypoxia. Pulmonary pressure and cardiac output will be measured during 60 minutes of poikilocapnic hypoxia.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years of age
* regularly physically active
* male

Exclusion Criteria:

* ex-smokers
* pulmonary function <80% of predicted
* contraindications to carbonic anhydrase inhibitors (eg. severe or absolute glaucoma, adrenocortical insufficiency, hepatic insufficiency, renal insufficiency, sulfa allergy or an electrolyte imbalance such as hyperchloremic acidosis)
* Obese (BMI>30Kg/m2)
* diuretic medication use
* blood thinner use
* anti-platelet drug use.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2016-05; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change in ventilation | Baseline and 60 minutes of poikilocapnic hypoxia
  To quantify the isocapnic hypoxic ventilatory response, the hypercapnic ventilatory response, and the hypercapnic hypoxic ventilatory response, ventilation will be measured throughout controlled changes in end-tidal gas levels. Each protocol will consist of 90s steps in end-tidal oxygen partial pressure from baseline through 65, 57, and 47 mmHg. For hypercapnic hypoxia, the end-tidal partial pressure for carbon dioxide will be increased from baseline to +6 mmHg for 7 minutes before reducing the end-tidal partial pressure of oxygen as above. The poikilocapnic hypoxic ventilatory response will be determined by measuring the change in ventilation from baseline throughout 60 minutes of poikilocapnic hypoxia (fraction of inspired oxygen = 0.12)
Change in pulmonary artery pressure | Baseline and 60 minutes of poikilocapnic hypoxia
  Pulmonary artery systolic pressure (PASP) will be derived using the modified Bernoulli equation and the regurgitant velocity across the tricuspid valve. Estimates of right atrial pressure will be evaluated based upon the collapsibility index of the inferior vena cave during a sniff test. The pulmonary artery pressure response will be measured during 60 minutes of exposure to poikilocapnic hypoxia (fraction of inspired oxygen = 0.12)

SECONDARY OUTCOMES:
Change in cerebral blood velocity | Baseline and 60 minutes
  To quantify the isocapnic hypoxic cerebral blood velocity response, the hypercapnic cerebral blood velocity response, and the hypercapnic hypoxic cerebral blood velocity response, cerebral blood velocity in the middle and posterior cerebral arteries will be measured throughout controlled changes in end-tidal gas levels. Each protocol will consist of 90s steps in end-tidal oxygen partial pressure from baseline through 65, 57, and 47 mmHg. For hypercapnic hypoxia, the end-tidal carbon dioxide partial pressure will be increased from baseline to +6 mmHg for 7 minutes before reducing the end-tidal oxygen partial pressure as above. The poikilocapnic hypoxic ventilatory response will be determined by measuring the change in ventilation from baseline throughout 60 minutes of poikilocapnic hypoxia (fraction of inspired oxygen = 0.12)

OTHER OUTCOMES:
change in arterial oxygen partial pressure | Baseline and 60 minutes
Change in arterial carbon dioxide partial pressure | Baseline and 60 minutes
Change in arterial pH | Baseline and 60 minutes
Change in heart rate | Baseline and 60 minutes
change in blood pressure | Baseline and 60 minutes
change in end-tidal oxygen and carbon dioxide partial pressure | Baseline and 60 minutes
Change in arterial oxygen saturation | Baseline and 60 minutes
Change in cardiac output | Baseline and 60 minutes of poikilocapnic hypoxia
  Cardiac output will be determined using the aortic time integral velocity and the diameter of the aortic valve annulus. Data will be collected at baseline and throughout exposure to poikilocapnic hypoxia (fraction of inspired oxygen = 0.12)
Change in pulmonary venous blood velocity | Baseline and 60 minutes of poikilocapnic hypoxia
  Doppler ultrasound will be used to measure the velocity of blood draining from the pulmonary vein at baseline and throughout exposure to poikilocapnic hypoxia (fraction of inspired oxygen = 0.12)
Hemoglobin | Baseline
albumin | Baseline
iron | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Glen E Foster, Ph.D., Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Kelowna, British Columbia, Canada